CLINICAL TRIAL: NCT03149289
Title: Treatment of Hepatitis C Virus Infection With Direct-acting Antiviral Drugs in Patients With Hemoglobinopathies
Brief Title: Hepatitis C Virus Infection in Patients With Hemoglobinopathies
Status: Completed | Type: Observational
Sponsor: Società Italiana Talassemie ed Emoglobinopatie (Other)
Collaborators: University of Cagliari (Other); University of Turin, Italy (Other); Azienda Ospedaliera Ospedali Riuniti Villa Sofia Cervello (Other); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other); Ente Ospedaliero Ospedali Galliera (Other); University of Campania Luigi Vanvitelli (Other); Cardarelli Hospital (Other); Reggio Calabria (Other); University of Palermo (Other)
Responsible Party: Sponsor
Other Study IDs: HCV-SITE
Record Dates: First submitted 2017-04-14; First posted 2017-05-11 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2017-01

CONDITIONS: Hepatitis C, Chronic; Hemoglobinopathies
MeSH Terms: conditions — Hepatitis C, Chronic; Hemoglobinopathies | interventions — Antiviral Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HCV RNA positive: hemoglobinopathies with hepatites C treated with antiviral drugs
  Interventions: Drug: Antiviral drugs

INTERVENTIONS:
Drug: Antiviral drugs — sofosbuvir, ribavirin, daclatasvir, ledipasvir, simeprevir, paritaprevir, dasabuvir, ombitasvir
  Other Names: Direct-acting antiviral drugs'

SUMMARY:
Progression of liver fibrosis in patients with hemoglobinopathies is strongly related to the severity of iron overload and the presence of chronic hepatitis C virus (HCV) infection. Effective iron chelation therapy and HCV infection eradication are efficacy to prevent liver complications. EASL and AASLD guidelines recommend interferon-free regimens for the treatment of HCV infection in patients with hemoglobinopathies. However, data regarding the use of direct-acting antiviral drugs (DAAs) in this patient population are very few This large, observational study evaluated the safety and efficacy of standard therapy with DAAs in a large Italian cohort of with hemoglobinopathies, chronic HCV infection and advanced liver fibrosis.

DETAILED DESCRIPTION:
Many patients with hemoglobinopathies have been infected with hepatitis C virus (HCV) through blood transfusion, mostly before screening of blood donors was introduced in 1992. The reported prevalence of anti-HCV-positive thalassemia patients varies between 4.4% in Turkey and 85.4% in Italy. HCV infection is associated with decompensated cirrhosis, hepatocellular carcinoma and other liver complications, especially if left untreated. Prevalence of cirrhosis in thalassemia patients up to 32% have been reported.

Thalassemia patients with cirrhosis have an increased risk of death. Progression of liver fibrosis is strongly related to the presence of chronic HCV infection and extent of iron overload. Thalassemia patients with elevated serum aminotransferase levels for >6 months should be tested for HCV infection and, in the event of HCV infection, HCV genotyping is recommended in order to plan antiviral therapy and the likelihood of response. Noninvasive transient elastography (FibroScan®) can be used to determine the presence of fibrosis in thalassemia patients with HCV infection.

Effective chelation therapy and treatment of HCV infection are needed in order to prevent liver complications and decrease morbidity and mortality. For many years, pegylated interferon (peg-IFN) plus ribavirin was the standard of care for the treatment of chronic HCV infection and decompensated cirrhosis. Studies of peg-IFN plus ribavirin have demonstrated sustained virological response (SVR) rates of 25-64% in patients with thalassemia and HCV infection. However, peg-IFN and ribavirin are both associated with anemia. Ribavirin-associated hemolysis leads to an increased requirement for blood transfusions, which in turn can lead to worsening of iron overload. Therefore, European Association for the Study of the Liver (EASL) 2015 guidelines recommend interferon-free regimens for the treatment of HCV infection in patients with hemoglobinopathies. The aim of this study was to evaluate the safety and efficacy of DAA standard regimens in patients with hemoglobinopathies and chronic HCV liver disease treated in Italy.

Antiviral treatments were administered according to Italian Medicines Agency (AIFA) guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hemoglobinopathies, chronic hepatitis due to HCV and the presence of fibrosis (defined as Fibroscan® stiffness ≥10 kPa) or a bioptic evaluation of cirrhosis (same ISHAK fibrosis score) determined within 6 months previously. Patients with extrahepatic manifestations of chronic hepatitis C virus infection (cryoglobulinemia with organ damage, B-lymphoproliferative disorders) were also included.

Exclusion Criteria:

* Patients with active cancer, including hepatocellular carcinoma, and pregnant or lactating females were excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with hemoglobinopathies with cronic hepatitis C
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2015-03-01; Primary Completion 2016-03-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Change in the number of participants with undetectable serum HCV RNA is being assessed at the end of treatment | baseline and 12 weeks
  The quantification of hepatitis virus particles in serum is assessed and expressed in IU/mL (IU, international units ) through quantitation of virus ribonucleic acid by real time polymerase chain reaction (PCR).

CONTACTS AND LOCATIONS:
Overall Officials: Vito Di Marco, MD, Study Director — University of Palermo, Palermo, Italy

IPD SHARING:
Plan to Share IPD: No